CLINICAL TRIAL: NCT01293305
Title: Randomized Evaluation Of Not Less Medical Association Chondroitin Sulfate Plus Glucosamine Sulfate (In Powder Dosage Forms And Oral Capsule), Manufactured By The Geolab Pharmaceutical Industry Ltd, Compared To The Drug Condroflex® (Powder And Oral Capsule), Manufactured In The Laboratory Zodiac, The Treatment Of Osteoarthritis.
Brief Title: Study With Chondroitin Sulfate and Glucosamine Sulfate (in Dosage Capsule and Sachet) in Treating Osteoarthritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azidus Brasil (Industry)
Responsible Party: Dr. Sergio Marcolino Rosa, LAL Clinica Pesquisa e Desenvolvimento Ltda.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CGSGEO1010
Record Dates: First submitted 2011-02-08; First posted 2011-02-10 (Estimated); Last update posted 2011-02-10 (Estimated); Status verified 2011-01

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Chondroitin Sulfates; Glucosamine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Chondroitin Sulfate + Glucosamine sulfate (Experimental): Pharmaceutical form capsule.
  Interventions: Drug: Chondroitin sulfate + Glucosamine sulfate
- Chondroitin Sulfate + Glucosamine Sulfate (Experimental): Oral powder.
  Interventions: Drug: Chondroitin sulfate + Glucosamine sulfate
- Condroflex® (Active Comparator): Pharmaceutical form capsule.
  Interventions: Drug: Chondroitin sulfate + Glucosamine sulfate
- CONDROFLEX® (Active Comparator): Oral powder
  Interventions: Drug: Chondroitin sulfate + Glucosamine sulfate

INTERVENTIONS:
Drug: Chondroitin sulfate + Glucosamine sulfate — 1 capsule three times daily, preferably in the same period
Drug: Chondroitin sulfate + Glucosamine sulfate — 1 sachet per day of the drug dissolved in a beaker with 200 mL water.

SUMMARY:
The use of chondroitin sulfate and glucosamine sulfate has been recognized since the 70 decade in the treatment of osteoarthritis. Numerous clinical trials have demonstrated the therapeutic properties of this association in control of osteoarthritis, especially in reducing pain and improving movement. The combination of chondroitin sulfate with glucosamine sulfate offers a significantly higher tolerance than most drug treatments and, moreover, has long lasting effects even after stopping treatment.

ELIGIBILITY:
Constitute the criteria for inclusion in the study:

* Patients who agree with all aspects of the study and sign the Informed Consent
* Patients older than 40 years, regardless of sex
* Patients with clinical and radiological osteoarthritis in at least one knee, grade 1, 2 or 3 (based on clinical and radiological criteria of Kellgren & Lawrence). In the case of involvement of both knees the knee will be evaluated with greater impairment due to illness
* Patients with symptoms of pain when moving the knee examined in the study on most days of the last month, also in view of randomization of study drugs (V0)
* Symptoms of osteoarthritis, expressed continuously or intermittently over the last 6 months preceding the study

Constitute the criteria for exclusion from the study:

* History of clinically significant trauma to less than 3 months and to keep the clinical signs of trauma
* Patients who have performed surgery (including arthroscopy) in the affected joints less than 3 months and, at the discretion of the investigators, might interfere with study evaluations
* clinical history compatible with arthropathy that may confuse or interfere with pain assessment and effectiveness, including an inflammatory arthropathy (rheumatoid arthritis, lupus erythematosus, espondialoartropatia, psoriatic arthritis, polymyalgia rheumatica) gout, episodes of acute monoarthritis consistent with pseudogout, Paget's disease with involvement of the joint study, a history of septic arthritis, and Wilson disease, hemochromatosis, alkaptonuria, primary osteochondromatosis, history of avascular necrosis or intra-articular fracture of the joint study
* Patients with isolated patellofemoral arthrosis
* Patients who are pregnant or of childbearing potential without contraception
* Patients who are breastfeeding
* Patients with a history of PKU
* Patients with clinical diagnosis of severe renal insufficiency
* Patients with clinical diagnosis of severe liver diseases
* Patients with clinical diagnosis of bleeding disorders
* Patients who are being treated with oral anticoagulants or systemic
* Treatment with corticosteroids:

Use of corticosteroids orally or intramuscularly, fast action, for up to two weeks before V-1 or 14 days before the scheduled visits Use of oral corticosteroids or intramuscular depot for up to 4 weeks before V-1 or 14 days before the scheduled visits the administration of intra-articular corticosteroids in the study joint in the 3 months prior to randomization visit (V0) or during the study the administration of intra-articular corticosteroid into any other joint for up to 4 weeks prior to randomization visit (V0) or during the study

* Patients who have received intra-articular injection of hyaluronic acid or counterparts in the joint study in the past 12 months and during the study period
* Topical use of analgesics and irregular in the joint under study (eg, capsaicin) due to the possibility of causing a worsening of pain
* Use oral and / or systemic analgesics high power (opioids, tramadol) often or last week before the inclusion visit (V0)
* Implementation of any other medical treatment for osteoarthritis in the month prior to entry in the trial or a change of medical treatment already available, such as aerobics or physical therapy
* Clinical diagnosis established uncontrolled diabetes mellitus, with fasting glucose greater than 126 mg / dL
* Patients with a history of daily consumption of alcohol or, at the discretion of the investigator, be considered abusive
* Patients with hypersensitivity or a history of clinical or laboratory adverse event to acetaminophen, chondroitin sulfate and glucosamine sulfate
* Patients with emotional disorders that interfere with the capture of data
* Patients who do not agree with the purposes of the study and did not sign the Informed Consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-08 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Promotion of pain relief in patients with osteoarthritis. | 4 months.
  Assessment of noninferiority clinical association Chondroitin + glucosamine in dosage forms and oral powder hard gelatin capsule, produced by Geolab Pharmaceutical Ltd., with the comparator drugs in the same dosage forms produced by the Laboratory Zodiac (Condroflex ®) through the promotion of pain relief in patients with osteoarthritis between grades 1 and 3, according to the classification of Kellgreen & Lawrence (1957), measured by visual analogue scale (VAS). There will be five visits: V0, V1, V2, V3 and V4.

SECONDARY OUTCOMES:
Functional capacity, overall assessment of clinical improvement, assessment of adverse events | 4 months.
  Are the secondary objectives:
  * Functional capacity before and after treatment, using the Lequesne questionnaire, comparing the groups (T and Co).
  * Overall evaluation of clinical improvement made by the principal investigator.
  * Incidence of use of painkillers and anti-inflammatory drugs orally for the treatment through the patient's report, comparing the groups (T and Co).
  * Evaluation of the incidence, type and intensity of adverse events during the study, comparing the groups (T and Co).